CLINICAL TRIAL: NCT07099521
Title: The Effects of High-definition Transcranial Direct Current Stimulation on Cognitive Bias Among Individuals With Social Anxiety Symptoms
Brief Title: The Effects of HD-tDCS on Cognitive Bias Among Individuals With Social Anxiety Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South China Normal University (Other)
Responsible Party: Principal Investigator, Yi Yu, Primary Investigator, South China Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCNU-PSY-2024-185
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS group (Active Comparator): Participants underwent 10 sessions of anodal (2mA, 20 minutes) HD-tDCS over 5 days targeting the left dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Active High-definition transcranial direct current stimulation
- Sham group (Sham Comparator): Participants underwent 10 sessions of sham HD-tDCS over 5 days targeting the left dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Sham high-definition transcranial direct current stimulation

INTERVENTIONS:
Device: Active High-definition transcranial direct current stimulation — Participants completed 10 sessions of anodal HD-tDCS stimulation over 5 consecutive days (two 20-minute sessions per day, with a 3-hour interval between sessions). Stimulation was delivered using an HD-tES device (Soterix Medical, Inc, Woodbridge, NJ, USA), targeting the left dorsolateral prefrontal context (DLPFC). In the active HD-tDCS condition, current was ramped up to 2mA over 30 seconds, maintained for 20 minutes, then ramped down to 0mA at the end.
  Arms: tDCS group
Device: Sham high-definition transcranial direct current stimulation — Participants completed 10 sessions of sham HD-tDCS stimulation over 5 consecutive days (two 20-minute sessions per day, with a 3-hour interval between sessions). Stimulation was delivered using an HD-tES device (Soterix Medical, Inc, Woodbridge, NJ, USA), targeting the left dorsolateral prefrontal context (DLPFC). In the sham condition, the current was ramped up to 2mA within the first and last 30 seconds to mimic the sensation of stimulation, but then ramped down, with no current maintained at other times.
  Arms: Sham group

SUMMARY:
To examine the offline effects of high-definition tDCS (HD-tDCS) on attention, interpretation and memory biases in youth with social anxiety.

DETAILED DESCRIPTION:
In current study, we adopted a comparative intervention study with randomized controlled in which we delivered multiple courses of offline anodal HD-tDCS over the left DLPFC. The aim of this study was to explore the offline impact of HD-tDCS on cognitive bias (including attention, interpretation and memory bias) among youth with social anxiety symptoms. In addition, the researchers sought to further investigate the impact of tDCS stimulation on social anxiety. We hypothesized that anodal tDCS would activates the left DLPFC to facilitate cognitive control of threat-related information among youth with social anxiety, thereby reducing threat attention, interpretation and memory bias, and even improving social anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 18 -24 years old
* No history of major organic brain diseases or mental disorders, and currently not taking hormone or mental disorder drugs, with no drug or alcohol dependence;
* No experience of transcranial direct current stimulation (tDCS) or transcranial magnetic stimulation (TMS) in the past six months;
* Participants are willing to participate and fill out the informed consent form;
* The score of the Patient Health Questionnaire (PHQ-9) is less than 5 points;
* The score of the Liebowitz Social Anxiety Scale (LSAS) is greater than or equal to 55 points

Exclusion Criteria:

* any psychiatric disorders;
* current or past diseases or injuries related to the brain;
* medical pumps, pacemakers and cochlear implants in the body;
* current pharmacological or mental treatments;
* tDCS or TMS experiences over past year were also excluded.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2024-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yu, Principal Investigator — South China Normal University; Yuanyuan Wang, Study Chair — South China Normal University
Locations (1):
- School of Psychology, South China Normal University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No
The original data will not be made public before the paper is published

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomly assigned to either tDCS or sham groups using a computer-generated randomization table, with a 1:1 allocation ratio. Participants remained blinded to treatment conditions throughout the intervention period. Researchers only received allocation information immediately prior to procedure implementation.
Groups:
- tDCS group: Participants underwent 10 sessions of anodal (2mA, 20 minutes) HD-tDCS over 5 days (2 times each day) targeting the left dorsolateral prefrontal cortex (DLPFC).
- Sham group: Participants underwent 10 sessions of sham HD-tDCS over 5 days (2 times each day) targeting the left dorsolateral prefrontal cortex (DLPFC).
Period: Overall Study
Arm/Group | tDCS group | Sham group
Started | 37 | 37
Completed | 34 | 32
Not Completed | 3 | 5
Not completed — Incompeleted stimulus program | 1 | 0
Not completed — Non-social anxiety symtpoms | 0 | 1
Not completed — Extreme values | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | tDCS Group | Sham Group | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Mean (Standard Deviation); unit: Number] | 20.62 (1.94) | 19.88 (1.91) | 20.26 (1.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 12 | 10 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han ethnicity | 32 | 32 | 64
  Others ethnicity | 2 | 0 | 2
Residence [Count of Participants; unit: Participants]
  Urban | 21 | 20 | 41
  Rural | 13 | 12 | 25
Only-child status [Count of Participants; unit: Participants]
  Yes | 13 | 10 | 23
  No | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Trial-level Bias Score (Negative)
Description: Assessment: Dot probe task;Indicator of Attention Avoidance. Dot probe task is a common experimental paradigm for measuring attention bias. After appearance of a fixed cross in the center of the computer screen, a pair of faces appear side by side. Then, a probe appears on the location previously occupied by one of the two faces. Participants were asked to response the location of the probe as quickly as possible and press the appropriate keys to answer.
  This study used the trail-level bias score (TL-BS) as a measure of the main outcomes of this task. TL-BS is an indicator of reaction time (RT), calculated by subtracting contiguous pairs of congruent trials (probe and emotional face appeared on the same location of the screen) from incongruent trials (probe and emotional face appeared on the opposite location of the screen).Negative scores represent avoidance of these stimuli. TL-BSnegative indicates the average value of TL-BSs <0ms
Time Frame: This task was administered at baseline (Day 1) and immediately after the last stimulation session (Day 5).
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | tDCS group | Sham group
Number analyzed (Participants) | 34 | 32
Milliseconds
  Pre-test | -54.92 (22.28) | -48.45 (17.96)
  Post-test | -44.29 (16.79) | -46.07 (18.71)

2. Primary Outcome: Endorsement Rates of Negative Interpretations
Description: Assessment: Word-sentence association paradigm; Indicator of Negative interpretation bias.
  Word sentence association paradigm (WSAP) was used to assess the interpretation bias in youth with social anxiety. Following the appearance of a fixed cross (500ms), an ambiguous sentence describing the social situation would be presented in the center of the screen (2000ms). Then, a word would appear at random for 500ms: the word might imply a threatening interpretation (e.g., "boring" or "rejection"), or imply a benign one (e.g., "captivating" or "accepted"). Participants were asked to decide whether the word was related to the ambiguous sentence ("F" for relevant and "J" for irrelevant).
  This study calculated the proportion of threaten interpretations that participants endorsed as being related to the sentence （Endorsement rates of negative interpretations）, which was prescribed as the primary result of interpretation bias.
Time Frame: This task was administered at baseline (Day 1) and immediately after the last stimulation session (Day 5)
Measure: Mean (Standard Deviation); unit: Proportion
Arm/Group | tDCS group | Sham group
Number analyzed (Participants) | 34 | 32
Proportion
  Pre-test | 0.48 (0.19) | 0.44 (0.18)
  Post-test | 0.41 (0.21) | 0.44 (0.22)

3. Secondary Outcome: Peak Trial-level Bias Score (Negative)
Description: Assessments: Dot-probe task; Indicator of Attention Avoidance. Dot probe task is a common experimental paradigm for measuring attention bias. After appearance of a fixed cross in the center of the computer screen, a pair of faces appear side by side. Then, a probe appears on the location previously occupied by one of the two faces. Participants were asked to response the location of the probe as quickly as possible and press the appropriate keys to answer.
  This study used the trail-level bias score (TL-BS) as a measure of the main outcomes of this task. TL-BS is an indicator of reaction time (RT), calculated by subtracting contiguous pairs of congruent trials (probe and emotional face appeared on the same location of the screen) from incongruent trials (probe and emotional face appeared on the opposite location of the screen).Negative scores represent avoidance of these stimuli. Peak TL-BSnegative indicates the minimum TL-BS value.
Time Frame: This task was administered at baseline (Day 1) and immediately after the last stimulation session (Day 5)
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | tDCS group | Sham group
Number analyzed (Participants) | 34 | 32
Milliseconds
  Pre-test | -189.32 (79.33) | -159.66 (86.08)
  Post-test | -133.09 (66.52) | -139.22 (62.64)

4. Secondary Outcome: Bias Score
Description: Assessments: Word-sentence association paradigm; Indicator of Negative interpretation bias.
  Word sentence association paradigm (WSAP) was used to assess the interpretation bias in youth with social anxiety. Following the appearance of a fixed cross (500ms), an ambiguous sentence describing the social situation would be presented in the center of the screen (2000ms). Then, a word would appear at random for 500ms: the word might imply a threatening interpretation (e.g., "boring" or "rejection"), or imply a benign one (e.g., "captivating" or "accepted"). Participants were asked to decide whether the word was related to the ambiguous sentence ("F" for relevant and "J" for irrelevant).
  This study recorded the response time and calculated the bias index (BI): threat BI = response times (reject threat - endorse threat) and benign BI = response times (endorse benign - reject benign).
Time Frame: This task was administered at baseline (Day 1) and immediately after the last stimulation session (Day 5)
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | tDCS group | Sham group
Number analyzed (Participants) | 34 | 32
Milliseconds
  Pre-test | -39.85 (383.45) | -92.98 (459.47)
  Post-test | -80.72 (363.52) | 45.72 (307.73)

5. Secondary Outcome: Recall Accuracy for Negative Words
Description: Assessments: free recall task; Indicator of negative memory bias. This study used free recall and recognition task to assess memory bias by the number of positive/negative words remembered. First, in the "encoding phase", after a short time for a fixed cross, words were presented randomly in turn . Participants were asked to read these words aloud and answer coding questions.After this phase, there was a 3-minute distraction task, during which participants were guided through 40 calculation problems. They were then given 2 minutes to freely recall the words that had appeared before, regardless of the order of the words. Next, they completed a recognition task. Recall Accuracy was calculated as: (number of correctly recall negative words) ÷ (total number of negative words presented).
Time Frame: This task was administered at baseline (Day 1) and immediately after the last stimulation session (Day 5)
Measure: Mean (Standard Deviation); unit: Proportion
Arm/Group | tDCS group | Sham group
Number analyzed (Participants) | 25 | 22
Proportion
  Pre-test | 0.15 (0.09) | 0.15 (0.08)
  Post-test | 0.13 (0.08) | 0.15 (0.09)

6. Secondary Outcome: Social Anxiety Symptoms
Description: Assessments: the Liebowitz Social Anxiety Scale. The Liebowitz Social Anxiety Scale (LSAS) was used to identify participants with social anxiety and to assess changes in social anxiety symptoms before and after the tDCS intervention. The scale contains 24 items, each of which assesses two aspects of fear and avoidance, using a 4-point Likert scale ("0" means "never" and "3" means "severe"), for a total of 48 items. A higher score indicated more severe social anxiety. The score ranges from 0 to 144. The total score would be categorized into 5 severity levels: 0-54 (normal), 55-64 (moderate), 65-79 (marked), 80-94 (severe), and ≥95 (very severe). In this study, participants scoring between 55 and 95 were included. The LSAS has demonstrated good internal consistency across three assessments (Cronbach's alpha = 0.87-0.90), and acceptable test-retest consistency (r = 0.47-0.79, p < 0.001).
Time Frame: Self-report questionnaires were administered at baseline (Day 1), immediately after the last stimulation session (Day 5), and at a 4-week follow-up (Day 30).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | tDCS group | Sham group
Number analyzed (Participants) | 33 | 31
Scores on a scale
  Pre-test | 72.7 (16.8) | 66.94 (12.72)
  Post-test | 63.39 (13.77) | 63.52 (13.89)
  Follow-up | 61.79 (12.09) | 60.42 (13.75)

7. Secondary Outcome: Trait Anxiety
Description: Assessments: the Spielberger Inventory - Trait (STAI-T). Trait anxiety was assessed using the Spielberger Trait Anxiety Inventory - Trait (STAI-T), which included 20 items rated on a 4-point scale, ranging from 20 to 80 (1 = "not at all" to 4 = "very much"). A higher score indicates severe trait anxiety symptoms. In this study, the STAI-T demonstrated good internal and test-retest reliability (Cronbach's alpha = 0.80-0.86; r = 0.69-0.79, p < 0.001).
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | tDCS group | Sham group
Number analyzed (Participants) | 33 | 31
Scores on a scale
  Pre-test | 39.74 (7.42) | 42.87 (5.95)
  Post-test | 36.55 (6.25) | 41.45 (7.40)
  Follow-up | 37.97 (7.65) | 42.03 (7.73)

8. Secondary Outcome: Negative Cognitive Bias (Attention Bias)
Description: Assessments: the Negative cognitive processing bias questionnaire; Indicator of self-report attention bias.
  Participants completed the Negative cognitive processing bias questionnaire (NCPBQ). The NCPBQ included 17 items divided into three subscales, along with three lie-detection items. Among it, the attention bias subscale includes 5 items (E.g., My attention is easily drawn to the tragic images on TV and is difficult to shift). Items were rated on a 5-point Likert scale from 1 ("disagree completely") to 5 ("agree completely"), with higher score indicating more severe cognitive bias. The score of attention bias subscale ranges from 5 to 25.
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | tDCS group | Sham group
Number analyzed (Participants) | 33 | 31
Scores on a scale
  Pre-test | 16.64 (4) | 15.81 (3.42)
  Post-test | 16.64 (4.20) | 15.58 (4.36)
  Follow-up | 16.12 (4.42) | 15.81 (4.48)

9. Primary Outcome: Recognition Accuracy for Negative Words
Description: Assessments: recognition task; Indicator of Negative Memory bias. This study used free recall and recognition task to assess memory bias by the number of positive/negative words remembered. First, in the "encoding phase", after a short time for a fixed cross, words were presented randomly in turn . Participants were asked to read these words aloud and answer coding questions.After this phase, there was a 3-minute distraction task, during which participants were guided through 40 calculation problems. They were then given 2 minutes to freely recall the words that had appeared before, regardless of the order of the words. Next, they completed a recognition task. Recognition Accuracy was calculated as: (number of correctly recognized negative words) ÷ (total number of negative words presented).
Time Frame: This task was administered at baseline (Day 1) and immediately after the last stimulation session (Day 5)
Population: Please note that a total of 47 participants completed the memory bias tasks (25 in the tDCS group, and 22 in the sham group).
Measure: Mean (Standard Deviation); unit: Proportion
Arm/Group | tDCS group | Sham group
Number analyzed (Participants) | 25 | 22
Proportion
  Pre-test | 0.84 (0.11) | 0.82 (0.13)
  Post-test | 0.77 (0.12) | 0.82 (0.16)

10. Secondary Outcome: Negative Cognitive Bias (Interpretation Bias)
Description: Assessments: the Negative cognitive processing bias questionnaire; Indicator of self-report interpretation bias.
  Participants completed the Negative cognitive processing bias questionnaire (NCPBQ). The NCPBQ included 17 items divided into three subscales, along with three lie-detection items. Among it, the interpretation bias subscale includes 5 items (E.g., If a new teacher is hard on me, I think it is because he sees me in a bad light and wants to get me in trouble). Items were rated on a 5-point Likert scale from 1 ("disagree completely") to 5 ("agree completely"), with higher score indicating more severe cognitive bias . The score of interpretation bias subscale ranges from 5 to 25.
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | tDCS group | Sham group
Number analyzed (Participants) | 33 | 31
Scores on a scale
  Pre-test | 15.39 (2.99) | 16.74 (3.43)
  Post-test | 15.36 (3.81) | 15.94 (4.40)
  Follow-up | 14.39 (3.97) | 15.81 (4.49)

11. Secondary Outcome: Negative Cognitive Bias (Memory Bias)
Description: Assessments: the Negative cognitive processing bias questionnaire; Indicator of self-report memory bias.
  Participants completed the Negative cognitive processing bias questionnaire (NCPBQ). The NCPBQ included 17 items divided into three subscales, along with three lie-detection items. Among it, the memory bias subscale includes 4 items (E.g., I can easily remember the negative comments people make about me). Items were rated on a 5-point Likert scale from 1 ("disagree completely") to 5 ("agree completely"), with higher score indicating more severe cognitive bias . The score of memory bias subscale ranges from 5 to 20.
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | tDCS group | Sham group
Number analyzed (Participants) | 33 | 31
Scores on a scale
  Pre-test | 16.06 (2.32) | 14.55 (2.22)
  Post-test | 16.09 (2.57) | 14.77 (2.79)
  Follow-up | 14.85 (3.38) | 14.52 (2.84)

ADVERSE EVENTS:
Time Frame: After each stimulation session, participants completed an adverse event checklist to monitor tolerability and perceived stimulation. In other words, every participant underwent adverse event assessments from the first to the last intervention, for up to five consecutive days.
Arm/Group | tDCS group | Sham group
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32
Other Adverse Events (participants affected / at risk) | 34/34 | 32/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | tDCS group (N=34) | Sham group (N=32)
Scalp pain (Skin and subcutaneous tissue disorders) | 24 | 27
Stabbing pain (Skin and subcutaneous tissue disorders) | 31 | 29
Itching (Skin and subcutaneous tissue disorders) | 19 | 17
Burning (Skin and subcutaneous tissue disorders) | 24 | 21
Skin redness (Skin and subcutaneous tissue disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT07099521/Prot_SAP_002.pdf
  • Informed Consent Form (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT07099521/ICF_003.pdf